CLINICAL TRIAL: NCT03123588
Title: A Double-Blind, Double-Dummy Phase 2 Randomized Study to Evaluate the Efficacy and Safety of Ruxolitinib Versus Anagrelide in Subjects With Essential Thrombocythemia Who Are Resistant to or Intolerant of Hydroxyurea (RESET-272)
Brief Title: Phase 2 Study of Ruxolitinib Versus Anagrelide in Subjects With Essential Thrombocythemia Who Are Resistant to or Intolerant of Hydroxyurea (RESET-272)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment issues
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-272 (RESET-272)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Essential thrombocythemia; hydroxyurea-resistant; hydroxyurea-intolerant; ruxolitinib; anagrelide
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential | interventions — ruxolitinib; anagrelide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A : Ruxolitinib and anagrelide placebo (Experimental): Ruxolitinib or placebo will be administered orally twice a day at a starting dose of 10 mg.
  Interventions: Drug: Ruxolitinib; Drug: Placebo
- Group B : Anagrelide and Ruxolitinib PLacebo (Active Comparator): Anagrelide or placebo will be administered orally twice a day at a starting dose of 1 mg. Use of anagrelide will be consistent with approved prescribing information.
  Interventions: Drug: Anagrelide; Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib administered orally twice daily (BID) at the protocol-defined starting dose.
  Other Names: Jakafi; INCB018424
  Arms: Group A : Ruxolitinib and anagrelide placebo
Drug: Anagrelide — Anagrelide administered orally at a starting dose of 1 mg BID.
  Arms: Group B : Anagrelide and Ruxolitinib PLacebo
Drug: Placebo — Anagrelide-placebo administered orally BID
  Arms: Group A : Ruxolitinib and anagrelide placebo
Drug: Placebo — Ruxolitinib-placebo administered orally BID.
  Arms: Group B : Anagrelide and Ruxolitinib PLacebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib versus anagrelide in subjects with essential thrombocythemia who are resistant to or intolerant of hydroxyurea.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of essential thrombocythemia according to revised World Health Organization (WHO) 2016 criteria.
* Resistant to or intolerant of hydroxyurea, that is, fulfilling at least 1 of the following criteria:

  * Platelet count > 600 × 10^9/L after 3 months of at least 2 g/day of hydroxyurea (2.5 g/day in subjects with a body weight over 80 kg) OR at the subject's maximally tolerated dose if that dose is < 2 g/day.
  * Platelet count > 400 × 10^9/L and WBC count < 2.5 × 10^9/L or hemoglobin < 10 g/dL at any dose of hydroxyurea.
  * Presence of leg ulcers or other unacceptable mucocutaneous manifestations at any dose of hydroxyurea.
  * Hydroxyurea-related fever.
* Platelet count ≥ 650 × 10^9/L at screening.
* WBC ≥ 11.0 × 10^9/L at screening.

Exclusion Criteria:

* Subjects previously treated with anagrelide or Hydroxyurea (HU).

  1. Prior anagrelide use is allowed provided the reason for discontinuation is not AE-related and anagrelide is stopped at least 28 days before the start of study medications (ie, Day 1).
  2. Treatment with HU can be stopped at any time once one of the inclusion criteria for HU refractoriness or resistance have been met, and up to the day before the first dose of study treatment (ie, Day 1).
* Inadequate liver function at screening and Day 1 (before drug administration) as demonstrated by:

  * Total bilirubin > 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase or alanine aminotransferase > 1.5 × ULN
  * Hepatocellular disease (eg, cirrhosis)
* Inadequate renal function at screening as demonstrated by creatinine clearance < 40 mL/min calculated by Cockcroft-Gault equation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, MD, Study Director — Incyte Corporation
Locations (26):
- United States (26):
  - Mayo Clinic, Phoenix, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - Innovative Clinical Research Institute, Whittier, California
  - Bond Clinic, PA, Winter Haven, Florida
  - Tift Regional, Tifton, Georgia
  - Edward Cancer Center, Naperville, Illinois
  - North Shore Cancer Research Association-Skokie, Skokie, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Clinical Trials of SWLA LLC, Lake Charles, Louisiana
  - St. Agnes Hospital, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Summit Medical Group, Morristown, New Jersey
  - Columbia Weill Cornell Cancer Centers - Herbert Irving Comprehensive Cancer Center (HICCC), New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Waverly Hem Onc, Cary, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Gabrail Cancer Center- Canton Facility, Canton, Ohio
  - INTEGRIS Southwest Medical Center, Oklahoma City, Oklahoma
  - INTEGRIS Cancer Institute Proton Campus, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Geisinger - Knapper Clinic, Danville, Pennsylvania
  - Prairie Lakes Health Care System Inc., Watertown, South Dakota
  - Renovatio Clinical, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 120 participants were planned for enrollment and 12 participants were enrolled (6 in the ruxolitinib group and 6 in the anagrelide group). The first participant was dosed on 14 Nov 2017 and Last participant completed study on 03 Aug 2020
Pre-assignment Details: Twelve participants were enrolled and randomized. One participant in the ruxolitinib group was enrolled in error and withdrawn from the study before receiving any dose of study drug.
Period: Overall Study
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib Placebo
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Study Terminated by Sponsor | 2 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (13.04) | 61.2 (16.77) | 66.5 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 5 | 6 | 11
  Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieve Platelet and White Blood Cell (WBC) Control
Description: Defined as proportion of subjects who achieve a simultaneous reduction of platelet counts to < 600 × 10^9/L with a reduction of WBC counts to < 10 × 10^9/L for at least 80% of biweekly measurements for a consecutive 12-week period between Weeks 32 and 52.
Time Frame: 52 weeks
Population: The intent-to-treat (ITT) population will include subjects randomized in the study
Measure: Number; unit: proportion of participants
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib PLacebo
Number analyzed (Participants) | 6 | 6
proportion of participants | 0 | 0.17

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Time Frame: Baseline through the end of randomized period -up to 14 months per participant
Population: The safety population includes all randomized subjects who received at least 1 dose of study drug. AE has been summarized only in randomized period. End of randomized period is defined as the earliest of discontinuation or the individual unblinding date.
Measure: Number; unit: participants
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib PLacebo
Number analyzed (Participants) | 5 | 6
participants | 5 | 4

3. Secondary Outcome: Proportion of Subjects Who Achieve Complete Remission or Partial Remission
Description: Defined as proportion of subjects who achieve CR or PR at Week 32 based on European LeukemiaNet (ELN) 2013 response criteria. Per ELN criteria: Complete Remission: durable resolution of disease related signs and symptoms, durable blood count normalization, absence of hemorrhagic or thrombotic events, absence of signs of progressive disease and bone marrow histological remission including disappearance of megakaryocyte hyperplasia and absence of reticulin fibrosis >Grade 1.
  Partial remission: durable resolution of disease related signs and symptoms, durable blood count normalization, absence of hemorrhagic or thrombotic events, absence of signs of progressive disease, persistance of megakaryocyte hyperplasia.
  No response: any response that does not satisfy partial remission. Progressive Disease: transformation in PET-MF, MDS or acute leukemia.
Time Frame: 32 weeks
Population: The intent-to-treat (ITT) population will include subjects randomized in the study
Measure: Number; unit: proportion of participants
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib Placebo
Number analyzed (Participants) | 6 | 6
proportion of participants | 0 | 0.17

4. Secondary Outcome: Time to Treatment Discontinuation
Description: Defined as the time when treatment is discontinued
Time Frame: 98 weeks
Population: The intent-to-treat (ITT) population will include subjects randomized in the study
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib Placebo
Number analyzed (Participants) | 5 | 6
Days | 261.2 (238.85) | 437.2 (183.99)

5. Secondary Outcome: Duration of Response
Description: Defined as measurement of response from the onset of response to the loss of response for responders.
Time Frame: 142 weeks
Population: The intent-to-treat (ITT) population who are responders
Measure: Number; unit: Days
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib PLacebo
Number analyzed (Participants) | 0 | 1
Days |  | 442

6. Secondary Outcome: Proportion of Subjects Who Achieve Reduction of Platelet Counts to < 600 × 10^9/L
Description: Defined as Proportion of subjects who achieve reduction of platelet counts to < 600 × 10^9/L for at least 80% of biweekly measurements for a consecutive 12-week period between Weeks 32 and 52.
Time Frame: Between 32 and 52 weeks
Population: The intent-to-treat (ITT) population will include subjects randomized in the study
Measure: Number; unit: Proportion of participants
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib Placebo
Number analyzed (Participants) | 5 | 6
Proportion of participants | 0 | 0.50

7. Secondary Outcome: Proportion of Subjects Who Achieve a Reduction of WBC Counts to < 10 × 109/L
Description: Defined as Proportion of subjects who achieve a reduction of WBC counts to < 10 × 109/L for at least 80% of biweekly measurements for a consecutive 12-week period between Weeks 32 and 52.
Time Frame: 52 weeks
Population: The intent-to-treat (ITT) population will include subjects randomized in the study
Measure: Number; unit: Proportion of participants
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib PLacebo
Number analyzed (Participants) | 5 | 6
Proportion of participants | 0 | 0.33

ADVERSE EVENTS:
Time Frame: Baseline through the end of randomized period -up to 14 months per participant
Description: The safety population includes all randomized subjects who received at least 1 dose of study drug. AE has been summarized only in randomized period. End of randomized period is defined as the earliest of discontinuation or the individual unblinding date.
Arm/Group | Group A : Ruxolitinib and Anagrelide Placebo | Group B : Anagrelide and Ruxolitinib Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A : Ruxolitinib and Anagrelide Placebo (N=5) | Group B : Anagrelide and Ruxolitinib Placebo (N=6)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A : Ruxolitinib and Anagrelide Placebo (N=5) | Group B : Anagrelide and Ruxolitinib Placebo (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood creatinine (Investigations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03123588/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT03123588/SAP_001.pdf